CLINICAL TRIAL: NCT02361710
Title: Comparing the Serum Vitamin D Levels and Pregnancy Rates in Women Undergoing Elective Frozen Embryo Transfer (eFET)
Brief Title: Serum Vitamin D Levels and Pregnancy Rates in Women Undergoing Elective Frozen Embryo Transfer (eFET)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bahceci Clinic (Other)
Responsible Party: Principal Investigator, C CELİK, Associate Professor, Bahceci Clinic
Other Study IDs: BHC24120209
Record Dates: First submitted 2015-02-08; First posted 2015-02-12 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Pregnancy
Keywords: Vitamin D; pregnancy rate; eFET

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- vitamin D deficient patients: Serum 25- (hydroxide) OH Vitamin D levels <20ng/L undergoing Frozen embryo transfer (Vitamin D levels are measured on the day of embryo transfer)
  Interventions: Procedure: frozen embryo transfer
- vitamin D sufficient patients: Serum 25- (hydroxide) OH Vitamin D levels >20ng/L undergoing Frozen embryo transfer (Vitamin D levels are measured on the day of embryo transfer)
  Interventions: Procedure: frozen embryo transfer

INTERVENTIONS:
Procedure: frozen embryo transfer — comparison of groups according to their serum vitamin D levels on frozen embryo transfer day

SUMMARY:
The aim of this study is determining the affects of serum vitamin D levels to implantation and clinical pregnancy rates in women undergoing elective vitrified/thawed embryo transfer. Two groups will be identified according to the serum vitamin D levels on eFET transfer day and later on implantation, clinical pregnancy and ongoing pregnancy rates will be compared between those groups

DETAILED DESCRIPTION:
In the last decade there have been growing evidence about Vitamin D receptors and their role in female genital tract. But these studies are yet not well designed and the results should be interpreted cautiously. Although some of these studies advocating the Vitamin D deficiency as an negative circumstance on pregnancy rates some of the others don't agree. According to contradictory results understanding the actual role of those receptors needs more observation.

Latest retrospective analyse postulated that, vitamin D deficiency in fresh single embryo transfer cycles may reduce pregnancy rates mediated by endometrium or ovarian reserve and stimulation characteristics.

For this reason the investigators aimed to explore the effect of serum Vitamin D levels on pregnancy rates in infertile population undergoing frozen embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 35 years age, a frozen ET with 1 Day 5 (blastocyst stage) embryo
* Infertile women undergoing ICSI (intracytoplasmic sperm injection) cycle
* Factors affecting fertility are Tubal
* Unexplained or ovulatory disturbances,

Exclusion Criteria:

* Need to do Preimplantation Genetic Diagnosis
* Presence of endometriosis and adenomyosis
* Severe male factor infertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women undergoing a frozen ET with 1 Day 5 (blastocyst stage) embryo
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks after embryo transfer
  The presence of intrauterine gestational sac at 7 weeks of gestation

SECONDARY OUTCOMES:
implantation rates | 3 weeks after embryo transfer
  number of gestational sacs per transferred embryo.
ongoing pregnancy rates | 18 weeks after embryo transfer
  Pregnancy that had completed ≥20 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: mustafa bahceci, Study Director — bahceci Fulya IVF center
Locations (1):
- Bahceci Fulya IVF Center, Istanbul, Fulya, Turkey (Türkiye)

REFERENCES:
- [Background] Rudick B, Ingles S, Chung K, Stanczyk F, Paulson R, Bendikson K. Characterizing the influence of vitamin D levels on IVF outcomes. Hum Reprod. 2012 Nov;27(11):3321-7. doi: 10.1093/humrep/des280. Epub 2012 Aug 21. PMID 22914766